CLINICAL TRIAL: NCT00447460
Title: A Phase I/II Trial in Treating Patients With Graft-Versus-Host Disease by the Infusion of Expanded in-Vitro Allogenic Mesenchymal Stem Cell
Brief Title: Treatment of Refractory (Acute or Chronic) Graft-Versus-Host Disease by the Infusion of Expanded in-Vitro Allogenic Mesenchymal Stem Cell
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Collaborators: Haematology Service,University Hospital of Salamanca, MªConsuelo del Cañizo Fernández-Roldán (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSM/EICH2005; EudraCT Number: 2005-003674-14
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2007-03-22 (Estimated); Status verified 2007-03

CONDITIONS: Graft-vs-Host Disease (GVHD)
Keywords: Graft-vs-host disease (GVHD); Mesenchymal stem cell (MSC); Allogeneic hematopoietic stem cell transplant; Allotransplant; Allogenic; Refractory; CSM/EICH2005
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Mesenchymal stem cell (MSC)

SUMMARY:
Clinical trial based on the use of a new therapeutic strategy (MSC infusion) for the treatment of patients who have developed a GVHD refractory to the usual therapeutic measures after undergoing an allogenic hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
This is a multicenter, single dose study of allogenic mesenchymal stem cell (1-2 x 10^6 MSC/Kg recipient´s bodyweight).

MSC will be infused, by a central venous catheter, to patients diagnosed with GVHD refractory to first-line or subsequent treatment.

All patients will receive the same treatment. MSC suspension will be obtained from the bone marrow aspiration of a family donor and expanded in-vitro in a specific culture medium with autologous donor´s serum and with no animal-derived products.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancies who had been undergone an allogenic hematopoietic stem cell transplant and diagnosed with GVHD refractory to a usual treatment.
* Adequate cardiac function with no evidence of uncontrolled high blood pressure,congestive heart failure, angina pectoris, acute myocardial infarction within 6 months prior to the process.
* Adequate pulmonary function with no evidence of chronic obstructive or severe restrictive pulmonary disease.
* Patients with ages between 18 and 65 years.
* Signature of informed consent form is required to be done by patient and donor.

Exclusion Criteria:

* Patients whose hematopathology has not been controlled by the transplant or is in progress.
* Patients with bacterial, viral or fungal infection not being controlled with the adequate treatment.
* Patients with an inadequate cardiac or pulmonary function.
* Patients who, in the investigator´s point of view, are not in situation to tolerate the treatment.
* Patients who do not have the required donor (HLA-identical sibling donor and not HLA-identical sibling donor).
* Pregnant females or childbearing potential who are not on adequate contraceptive measures.
* Patients <18 or >65 years.
* Patients who do not sign the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2007-01; Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Determine the safety/efficacy of expanded in-vitro allogenic mesenchymal stem cell infusion in patients developing a GVHD refractory to the usual therapeutic measures after undergoing an allogeneic hematopoietic stem cell transplant.
Efficacy will be evaluated in terms of GVHD response.
Safety will be evaluated in terms of incidence of adverse events and toxicities related to the administration of MSC.

SECONDARY OUTCOMES:
Evaluation of infectious complications after MSC infusion.
Analyse the influence of MSC infusion on the posttransplant relapse risk of the base disease.
Study the influence of MSC infusion on DFS and OS.
Determine MSC grafted into the bone marrow (or in other organs).

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo del Cañizo, MD, Study Chair — Haematology Service, University Hospital of Salamanca; José A Pérez-Simón, MD, Principal Investigator — Haematology Service, University Hospital of Salamanca; David Varcárcel Ferrerías, MD, Principal Investigator — Haematology Service, Santa Creu i Sant Pau Hospital, Barcelona; Carmen Martínez Muñoz, MD, Principal Investigator — Haematology Service, Clinic i Provincial Hospital, Barcelona; José Rifón Roca, MD, Principal Investigator — Haematology Service, University Clinic of Navarra
Locations (4):
- Spain (4):
  - Santa Creu i Sant Pau Hospital, Barcelona, Barcelona
  - Clinic i Provincial Hospital, Barcelona, Barcelona
  - University Clinic of Navarra, Navarra, Pamplona
  - University Hospital of Salamanca, Salamanca, Salamanca

REFERENCES:
- [Derived] Perez-Simon JA, Lopez-Villar O, Andreu EJ, Rifon J, Muntion S, Diez Campelo M, Sanchez-Guijo FM, Martinez C, Valcarcel D, Canizo CD. Mesenchymal stem cells expanded in vitro with human serum for the treatment of acute and chronic graft-versus-host disease: results of a phase I/II clinical trial. Haematologica. 2011 Jul;96(7):1072-6. doi: 10.3324/haematol.2010.038356. Epub 2011 Mar 10. PMID 21393326